CLINICAL TRIAL: NCT00853333
Title: Sedation and Pain (The Effect of IV Sedation on Pain Perception)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Society of Regional Anesthesia (Other)
Responsible Party: Principal Investigator, Michael Froelich, M.D., University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: F081016014
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: Pain; Propofol; Dexmedetomidine; Midazolam; Effects of sedation on pain perception.
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Midazolam; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Propofol (Active Comparator): Administration via an IV
  Interventions: Drug: propofol
- Midazolam (Active Comparator): Administration via an IV
  Interventions: Drug: midazolam
- Dexmedetomidine (Active Comparator): Administration via an IV
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine
  Arms: Dexmedetomidine
Drug: midazolam
  Arms: Midazolam
Drug: propofol
  Arms: Propofol

SUMMARY:
The investigators propose to evaluate the potential effect of sedation on pain perception in two ways, by asking for a participant's pain rating(subjective) and by evaluating a subject's brain activation using fMRI(objective).

DETAILED DESCRIPTION:
We propose to contrast and compare the effect of propofol and midazolam, two GABA-related sedative drugs, and dexmedetomidine, an alpha-2 adrenergic agonist, on pain perception in human volunteers by asking a participant to rate their pain and by evaluating a subject's brain activation using fMRI.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects

* 19 years or older able to follow study instructions

Exclusion Criteria:

* Age less than 19 or greater than 40
* Pregnant female
* Obesity (BMI > or =35)
* Non-English speaking/reading participants
* Sleep apnea
* Pulmonary problems such as moderate or severe bronchial asthma
* Cardiovascular problems such as hypertension
* History of claustrophobia
* Presence of a pacemaker, defibrillator, surgically placed metallic object (e.g., hip replacement)or other implanted device
* Presence of an unremoved bullet or shrapnel in the body
* Presence of a prosthetic that is not removable
* Presence of a hearing aid needed for hearing
* Head girth exceeding that of the head coil used in the magnet
* Extensive metalwork on or in teeth, or irremovable false teeth or bridgework
* Epilepsy
* Chronic analgesic medication
* Excessive tattoos (due to local skin heating with tattoos containing ferromagnetic particles)
* History of surgery for which details are unavailable
* Allery due to study drugs
* History of drug abuse

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2008-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Froelich, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Frolich MA, Zhang K, Ness TJ. Effect of sedation on pain perception. Anesthesiology. 2013 Mar;118(3):611-21. doi: 10.1097/ALN.0b013e318281592d. PMID 23314164

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine: Sedation Arm 1, Dose adjusted to Sedation Self-rating of 50% on Sedation Scale.
- Midazolam: Sedation Arm 2, Dose adjusted to Sedation Self-rating of 50% on Sedation Scale.
- Propofol: Sedation Arm 3, Dose adjusted to Sedation Self-rating of 50% on Sedation Scale.
Period: Overall Study
Arm/Group | Dexmedetomidine | Midazolam | Propofol
Started | 28 | 27 | 31
Completed | 28 | 27 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Midazolam | Propofol | Total
Number analyzed (Participants) | 28 | 27 | 31 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.74 (4.47) | 24.46 (4.64) | 25.83 (5.41) | 25.01 (4.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 14 | 45
  Male | 13 | 11 | 17 | 41
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 31 | 86

OUTCOME MEASURES:

1. Primary Outcome: Pain Rating Change
Description: Mechanical Slide Algometer (www.decisionaidsonline.com), Range: "No Pain Sensation" (1) to " Most Intense Sensation Imaginable" (10) 10 point scale.
  Change Time Points: Baseline (no sedation), Sedation. Same Day Intervention.
Time Frame: Sedation
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Dexmedetomidine | Midazolam | Propofol
Number analyzed (Participants) | 28 | 27 | 31
units on a scale | -0.253 (0.168) | 0.762 (0.171) | -0.346 (0.159)

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine | Midazolam | Propofol
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/31
Other Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No